CLINICAL TRIAL: NCT03669757
Title: A Phase 1b, Randomised, Controlled, Observer-blinded Trial to Assess Safety, Tolerability and Pharmacodynamic Effects of LEO 134310 Cutaneous Solution in Descaled Skin of Adults With Chronic Plaque Psoriasis
Brief Title: Clinical Trial to Assess Safety, Tolerability and the Pharmacodynamic Effect of Different Concentrations of a New Anti-inflammatory Substance in Subjects With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP0155-1375; 2018-000140-26 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-09-13 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2019-02

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison of all treatment
Who Masked: Investigator
Masking Description: The trial will be performed investigator-blind with random assignment of the 4 Investigational Medicinal Products (IMPs), the placebo and the active comparator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- LEO 134310 Dose A (Experimental): Once daily application
  Interventions: Drug: LEO 134310
- LEO 134310 Dose B (Experimental): Once daily application
  Interventions: Drug: LEO 134310
- LEO 134310 Dose C (Experimental): Once daily application
  Interventions: Drug: LEO 134310
- LEO 134310 Dose D (Experimental): Once daily application
  Interventions: Drug: LEO 134310
- LEO 134310 vehicle (Placebo Comparator): Once daily application
  Interventions: Drug: LEO 134310 vehicle
- 0.1% betamethasone valerate ointment (class III steroid) (Active Comparator): Once daily application
  Interventions: Drug: 0.1% betamethasone valerate ointment (class III steroid)

INTERVENTIONS:
Drug: LEO 134310 — Active substance: LEO 134310 is a compound in development at LEO Pharma A/S
  Arms: LEO 134310 Dose A
Drug: LEO 134310 — Active substance: LEO 134310 is a compound in development at LEO Pharma A/S
  Arms: LEO 134310 Dose B
Drug: LEO 134310 — Active substance: LEO 134310 is a compound in development at LEO Pharma A/S
  Arms: LEO 134310 Dose C
Drug: LEO 134310 — Active substance: LEO 134310 is a compound in development at LEO Pharma A/S
  Arms: LEO 134310 Dose D
Drug: LEO 134310 vehicle — Active substance: none
  Arms: LEO 134310 vehicle
Drug: 0.1% betamethasone valerate ointment (class III steroid) — Active substance: betamethasone valerate
  Arms: 0.1% betamethasone valerate ointment (class III steroid)

SUMMARY:
To assess safety and tolerability after treatment with LEO 134310 cutaneous solution.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-64 years (inclusive) with plaque psoriasis in a chronic stable phase.
* Men or women of non-child bearing potential.

Exclusion Criteria:

* Acute psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica, pustular, exfoliative or inverse psoriasis.
* According to defined washout periods: topical antipsoriatic drugs (except salicylic acid in petroleum jelly); systemic antipsoriatics and biologics; ultraviolet (UV) therapy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Overall number of treatment-emergent adverse events. | Up to Day 19
Number of treatment-emergent application site reactions, by treatment. | Up to Day 19
Change from baseline to Day 4, Day 8 and Day 12 in haematology parameters | Up to Day 12
  red blood cells, white blood cells, hemoglobin, hematocrit, MCH, MMCV, MCHC, platelets, white cell differentials, measure in SI units
Change from baseline to Day 4, Day 8 and Day 12 in clinical chemistry parameters | Up to Day 12
  sodium, potassium, chloride, bicarbonate, blood urea nitrogen, glucose, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gammaGT, uric acid, calcium, phosphate, albumin, triglycerides, cholesterol, lactate dehydrogenase, total protein, creatinine, total bilirubin, direct bilirubin, indirect bilirubin
Change from baseline to Day 4, Day 8 and Day 12 in urinalysis parameters | Up to Day 12
  Single parameters only to be listed if deviation from usual urine dip test, e.g., sediment, leucocytes, nitrite, pH, protein, glucose, ketones, urobilinogen, bilirubin, blood/haemoglobin
Number of subjects with abnormal clinical significant ECG evaluation | Up to Day 12
  Evaluation of 12-lead ECG (overall evaluation, assessed by investigator as 'normal', 'abnormal not clinically significant', 'abnormal clinically significant')
Number of subjects with abnormal clinically significant findings of physical examination at Day 12. | Up to Day 12
  Evaluation of physical examination (areas skin, heart, lung, abdomen, basic neurological status, general examination of eyes, ears, nose throat), overall evaluation, assessed by investigator as 'normal', 'abnormal not clinically significant', 'abnormal clinically significant'
Change from baseline to Day 4, Day 8, Day 12 in systolic and diastolic blood pressure. | Up to Day 12
  measured in mmHg
Change from baseline to Day 4, Day 8 and Day 12 in pulse. | Up to Day 12
  measured in beats per minute
Change from baseline to Day 4, Day 8 and Day 12 in oral body temperature. | Up to Day 12
  measured in degrees celsius

SECONDARY OUTCOMES:
Change from baseline to Day 4, Day 8 and Day 12 in psoriatic infiltrate thickness (assessed by measurement of the thickness of the Echo Poor Band [EPB] of the inflammatory infiltrate using 22-MHz sonography) | 12 days
Change from baseline to Day 12 in disease severity | 12 days
  Clinical assessment of change in disease severity (a global assessment performed by an investigator using a 5-point score ('-1 = worsened', '0 = unchanged', '1 = slight improvement', '2 = clear improvement but not completely healed', '3 = completely healed')

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — LEO Pharma
Locations (2):
- Germany (2):
  - Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: No